CLINICAL TRIAL: NCT00645528
Title: Do Group Insulin Education Visits Reduce Barriers to Insulin Initiation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SHP 08-198
Record Dates: First submitted 2008-03-21; First posted 2008-03-27 (Estimated); Results first posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: insulin; teaching
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin Education Class Participants (Experimental): Participation in an insulin educational class at week 0 and again at week 2
  Interventions: Other: Insulin Education Class

INTERVENTIONS:
Other: Insulin Education Class — Participation in an Insulin Education Class at week 0 and week 2

SUMMARY:
The purpose of this research is to determine if meeting in a group with other subjects with diabetes can reduce barriers to starting insulin.

DETAILED DESCRIPTION:
Diabetes is a common, morbid and expensive disease among veterans. Achieving and maintaining adequate glycemic control can reduce the devastating complications of diabetes. Unfortunately a large percentage of veterans with type 2 diabetes continue to have poorly controlled blood sugars. Insulin is the most potent medication for reducing glycemia, but is not used often enough due to barriers that are both patient and provider driven.

We propose to conduct a pilot study to evaluate the feasibility of establishing an insulin education group that would serve to educate patients about insulin, to initiate insulin in a group setting, and to provide appropriate follow-up of those who start insulin. If the intervention is successful, we plan to develop a multicenter study to test rigorously the effect of this approach.

Specific Aims:

To determine if psychological barriers to insulin initiation in patients with uncontrolled type 2 diabetes are favorably affected by a group insulin education and insulin initiation visit, as measured by the Barriers to Insulin Treatment (BIT) Questionaire before and after the intervention.

To evaluate the feasibility of the intervention as measured by the percent of patients who are referred to the class, but either cancel without rescheduling or fail to report and the percent of patients who begin insulin.

To evaluate the safety of the intervention as measured by the proportion of patients experiencing hypoglycemic symptoms; proportion of patients requiring sugar intake to manage hypoglycemia; and the proportion of patients requiring assistance to manage hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Primary care patient at McGuire Veterans Affairs Medical Center in Richmond, Virginia
* Age > 18 years
* Inadequately controlled diabetes (HbA1c > 8.0%) and not on insulin (using most recent HbA1c, within 1 month of the first visit)
* Primary Care Provider referral to insulin initiation/education group
* Patient brings home glucose readings to first visit

Exclusion Criteria:

* Patient is reluctant to participate in a group visit for any reason
* Patient unwilling to sign consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonja K Fredrickson, MD, Principal Investigator — Hunter Holmes McGuire VA Medical Center
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were referred by their primary care provider (PCP) through an electronic consult to participate in an insulin education and initiation group visit. All patients received the same education and standard of care; however, only those subjects who signed an informed consent form and met inclusion/exclusion criteria had their data analyzed.
Pre-assignment Details: From April to July 2008, 102 patients were referred to the clinic, and 71 (70%) reported to visit 1. Of these, 32 were excluded: 15 did not bring a glucose log; 7 had HbA1c <8; 1 did not have HbA1c within 1 month; 1 was not referred by PCP; 6 did not consent; 2 were already on insulin. 39 were eligible for the study. 32 completed the study.
Groups:
- Insulin Education Class Participants: Subjects attended two group visits, two weeks apart, during which they received education regarding goals of therapy, insulin use, and hypoglycemia. Self-monitored blood glucose values were reviewed and insulin was initiated, if felt appropriate by the physician investigator and if accepted by the subject. The Barriers to Insulin Treatment Questionnaire (BIT) was completed at the start of the first visit and at the end of the second visit.The BIT is a 14 item self-administered questionnaire with 5 subscales, each representing a different psychological barrier to insulin treatment.
  Additionally, at the second visit, proportion of blood glucose readings below 70 mg/dl were recorded. All patients were asked how many times in the two weeks they experienced symptoms/signs of low blood sugar, how many times they required sugar intake for the these symptoms, and how many times they required another person to assist them.
Period: Overall Study
Arm/Group | Insulin Education Class Participants
Started | 39
Completed | 32
Not Completed | 7
Not completed — Did not show up for Visit 2 | 7

BASELINE CHARACTERISTICS:
Population: Subjects were eligible to participate if they (a) were referred to the group by their primary care provider; (b) had uncontrolled diabetes (hemoglobin A1c (A1c) >= 8.0%) not treated with insulin; (c) brought a glucose log to the first visit and (d) signed a consent form.
Groups:
- Insulin Education Class Participants: Participation in an insulin educational class
  Group Education: Participation in an insulin educational class
Arm/Group | Insulin Education Class Participants
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in "Barriers to Insulin Treatment (BIT)" Score From Before to After the Classes
Description: The Barriers to Insulin Treatment Questionnaire (BIT) was completed at the start of the first visit and at the end of the second visit. The BIT is a 14 item self-administered questionnaire with 5 subscales, each representing a different psychological barrier to insulin treatment. Scales are scored 1-10, representing the mean answer of the 10-point Likert questions for the relevant scale. The higher the score, the greater the barriers to insulin treatment, with the exception of the 2nd scale ("Expectations regarding positive insulin-related outcomes") where the lower the score, the greater the barriers to insulin treatment. An overall sum score is calculated the same way, after inverting the items of the 2nd scale. The overall sum scale is scored 1-10, representing the mean answers of the 10-point Likert questions. The higher the score, the greater the barriers to insulin treatment. Reported here is the change in BIT score from baseline. This was assessed by paired t-test.
Time Frame: 2 weeks
Population: 32 subjects completed the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Insulin Education Class Participants
Number analyzed (Participants) | 32
units on a scale
  Change in Total Sum Score | -0.76 (1.46)
  Change in Fear of Injections and Self-Testing | -0.42 (2.95)
  Change in Expectations regarding positive insulin | 0.88 (2.44)
  Change in Expected hardship from insulin therapy | -0.55 (2.62)
  Change in Stigmatization by insulin injections | -1.1 (2.33)
  Change in Fear of hypoglycemia | -1.02 (3.44)

2. Secondary Outcome: Percent of Patients Who Begin Insulin
Time Frame: 2 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Education Class Participants
Number analyzed (Participants) | 32
percentage of participants | 78

3. Secondary Outcome: Number of Subjects Experiencing Hypoglycemic Symptoms
Description: Number of subjects who reported subjective symptoms of hypoglycemia in the two weeks between study visits
Time Frame: 2 weeks
Population: As below, 15 subjects reported subjective symptoms of hypoglycemia in the two weeks between study visits; 10 of these subjects had at least one recorded blood glucose value less than 70 mg/dl; Eight of these 10 subjects had started insulin.
Measure: Number; unit: participants
Arm/Group | Insulin Education Class Participants
Number analyzed (Participants) | 32
participants | 15

4. Secondary Outcome: Number of Patients Experiencing a Severe Hypoglycemic Event
Description: Severe hypoglycemia is defined as requiring the help of another person to treat the hypoglycemia
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Insulin Education Class Participants
Number analyzed (Participants) | 32
participants | 0

5. Primary Outcome: Barriers to Insulin Treatment Total Sum Score Visit 1 (Week 0)
Description: The Barriers to Insulin Treatment Questionnaire (BIT) was completed at the start of the first visit and at the end of the second visit. The BIT is a 14 item self-administered questionnaire with 5 subscales, each representing a different psychological barrier to insulin treatment. Scales are scored 1-10, representing the mean answer of the 10 point Likert questions for the relevant scale. The higher the score, the greater the barriers to insulin treatment, with the exception of the 2nd scale ("Expectations regarding positive insulin-related outcomes") where the lower the score, the greater the barriers to insulin treatment. An overall sum score can be calculated the same way, after inverting the items of the 2nd scale. The overall sum scale is scored 1-10, representing the mean answers of the 10-point Likert questions. The higher the score, the greater the barriers to insulin treatment. The Total Sum Score and each subscale at Visit 1 is reported here.
Time Frame: Visit 1 (week 0)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Insulin Education Class Participants
Number analyzed (Participants) | 32
units on a scale
  Total Sum Score | 4.27 (1.29)
  Fear of injections and self-testing | 3.06 (2.24)
  Expectations regarding positive insulin-related ou | 5.59 (2.31)
  Expected hardship from insulin therapy | 4.16 (2.12)
  Stigmatization by insulin injections | 4.14 (1.74)
  Fear of hypoglycemia | 4.69 (2.62)

6. Primary Outcome: Barriers to Insulin Treatment Total Sum Score Visit 2 (Week 2)
Description: The Barriers to Insulin Treatment Questionnaire (BIT) was completed at the start of the first visit and at the end of the second visit. The BIT is a 14 item self-administered questionnaire with 5 subscales, each representing a different psychological barrier to insulin treatment. Scales are scored 1-10, representing the mean answer of the 10-point Likert questions for the relevant scale. The higher the score, the greater the barriers to insulin treatment, with the exception of the 2nd scale ("Expectations regarding positive insulin-related outcomes") where the lower the score, the greater the barriers to insulin treatment. An overall sum score is calculated the same way, after inverting the items of the 2nd scale. The overall sum scale is scored 1-10, representing the mean answers of the 10-point Likert questions. The higher the score, the greater the barriers to insulin treatment. The Total Sum Score and each subscale at Visit 2 is reported here.
Time Frame: Visit 2 (week 2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Insulin Education Class Participants
Number analyzed (Participants) | 32
units on a scale
  Total Sum Score | 3.51 (1.41)
  Fear of injections and self-testing | 2.64 (2.30)
  Expectations regarding positive insulin-related ou | 6.47 (1.84)
  Expected hardship from insulin therapy | 3.61 (2.29)
  Stigmatization by insulin injections | 3.13 (2.00)
  Fear of hypoglycemia | 3.79 (2.24)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at Visit 2, which occurred 2 weeks after Visit 1.
Groups:
- Arm 1: Participation in an insulin educational class
  Group Education: Participation in an insulin educational class
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 15/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=32)
Subjective Symptoms of hypoglycemia (Endocrine disorders) | 15
Recorded blood glucose less than 70 mg/dl (Endocrine disorders) | 10

LIMITATIONS AND CAVEATS:
This was a pilot study. Limitations include the small sample size and lack of a control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes